CLINICAL TRIAL: NCT07027748
Title: Feasibility Study of Prolonged Administration of Naxitamab, Irinotecan, and Temozolomide for Patients With Relapsed or Refractory Neuroblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Steven DuBois, MD (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Steven DuBois, MD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-211
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma; Neuroblastoma Recurrent; Relapsed Neuroblastoma; Refractory Neuroblastoma
Keywords: Neuroblastoma; Neuroblastoma Recurrent; Relapsed Neuroblastoma; Refractory Neuroblastoma; Progressive Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab; Irinotecan; Temozolomide; sargramostim

STUDY DESIGN:
Intervention Model Description: Participants are enrolled sequentially into cohorts corresponding to different naxitamab infusion durations and following a modified 3+3 design for safety assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Naxitamab Infusion+ Ironotecan + Temozolomide + Sargramostim (Experimental): Participants will be enrolled in a modified 3+3 design to establish a maximum tolerated, infusion duration for Naxitamab. Dosage will start at Duration Level 1 and will de-escalate to Duration Level -1 or escalate to Duration Level 2 according to dose-limiting toxicity (DLT) criteria.
  * Baseline visit
  * Cycle 1 (21 day cycle):
    * Days 1, 3, and 5: Predetermined dose of Naxitamab 1x daily
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 through 5: Predetermined dose of Ironotecan 1x daily
    * Days 6 through 12: predetermined dose of Sargramostim 1x daily
  * Cycles 2 through 6 (21 day cycles):
  * Imaging on Cycles 2, 4, and 6
    * Days 1, 3, and 5: Predetermined dose of Naxitamab 1x daily
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 through 5: Predetermined dose of Ironotecan 1x daily
    * Days 6 through 12: predetermined dose of Sargramostim 1x daily
  * End of treatment visit
  * Follow up at 1 year post-treatment
  Interventions: Drug: Naxitamab; Drug: Irinotecan; Drug: Temozolomide; Drug: Sargramostim granulocyte-macrophage colony stimulating factor

INTERVENTIONS:
Drug: Naxitamab — Recombinant humanized anti-GD2 monoclonal antibody, single-use vial, via intravenous (into the vein) infusion per protocol.
Drug: Irinotecan — Topoisomerase Inhibitor, single-dose vial, via intravenous infusion per standard of care
Drug: Temozolomide — Alkylating agent, capsule, via orally (by mouth) per standard of care
  Other Names: Temodal; Temodar
Drug: Sargramostim granulocyte-macrophage colony stimulating factor — Recombinant human granulocyte-macrophage colony stimulating factor (rhu GM-CSF), multi-use vial, via subcutaneously (under the skin) injection per standard of care
  Other Names: Leukine

SUMMARY:
This research is being done to investigate a treatment regimen of Irinotecan, Temozolomide, and Sargramostin, and an immunotherapy called Naxitamab and whether giving Naxitamab more slowly reduces the side effects for participants with relapsed or refractory neuroblastoma.

The name of the study drugs involved in this study are:

* Naxitamab (A type of monoclonal antibody)
* Irinotecan (A standard of care chemotherapy)
* Temozolomide (A standard of care chemotherapy)
* Sargramostim (A standard of care, granulocyte-macrophage colony stimulating factor)

DETAILED DESCRIPTION:
This phase 1, single treatment arm, prospective trial is designed to identify the maximally safe infusion duration of Naxitamab in combination with Irinotecan, Sargramostim, and Temozolomide for participants with relapsed, refractory, progressive neuroblastoma. Study doctors are studying different Naxitamab infusion duration levels (how quickly the drug is given into the vein) to determine if this makes a difference in side effects such as pain or infusion reactions.

Not every participant in this research study will receive the same infusion duration of the study drug, Naxitamab. The infusion duration received will depend on the number of participants who have been enrolled in the study and how well an infusion duration is tolerated.

The duration groups will be as follows:

* Duration Level -1: Naxitamab infusion duration will be 5 hours
* Duration Level 1: Naxitamab infusion duration will be 4 hours
* Duration Level 2: Naxitamab infusion duration will be 3 hours

The U.S. Food and Drug Administration (FDA) has approved Naxitamab for patients aged greater than 1 year with relapsed/refractory neuroblastoma in the bone or bone marrow.

The research study procedures include screening for eligibility, in-clinic visits, questionnaires, blood tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Meta-Iodine odobenzylguanidine (MIBG) scans, echocardiograms (ECGs), bone marrow aspiration/biopsies.

It is expected that about 18 people will take part in this research study.

YmAbs Therapeutics is supporting this research study by providing naxitamab for the trial and support to measure naxitamab blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Histologic Diagnosis: Patients must have had histologic verification of neuroblastoma or ganglioneuroblastoma or demonstration of neuroblastoma cells in the bone marrow with elevated urinary catecholamines [i.e. > 2 x upper limit of normal (ULN)], at the time of initial diagnosis.
* Relapsed or Refractory Disease Patients must have ONE of the following:

  * 1) Any prior episode of recurrent high-risk disease following completion of frontline high-risk therapy. Patients may have received other lines of therapy for treatment of recurrent disease prior to enrolling to this trial.
  * 2) Prior progressive high-risk disease during frontline high-risk therapy. Patients may have received other lines of therapy for treatment of progressive disease prior to enrolling to this trial.
  * 3) Primary resistant/refractory disease (less than partial response by INRC) detected after the conclusion of at least 4 cycles of aggressive multidrug induction chemotherapy on or according to a high-risk neuroblastoma protocol (examples include ANBL0532, ANBL09P1, ANBL12P1, ANBL1531, ANBL2131) that was treated with additional therapy with the goal of improving remission status prior to enrolling to this trial.
* Documentation of Disease: Patients must have at least ONE of the following at the time of enrollment:

  * 1) Measurable tumor on MRI or CT scan. Measurable is defined as ≥ 10 mm in at least one dimension (or 15 mm in short axis for lymph node) on spiral/helical CT or MRI that is MIBG avid or demonstrates increased FDG uptake on PET scan.
  * 2) MIBG-avid lesion detected on MIBG scan with positive uptake at a minimum of one site. This site must represent disease recurrence or known refractory disease at a site not previously radiated.
  * 3) In patients with known MIBG non-avid disease, FDG-avid lesion detected on FDG- PET scan with positive uptake at a minimum of one site. This site must represent disease recurrence or known refractory disease at a site not previously radiated.
  * Of note, patients with isolated bone marrow only disease are NOT eligible for this trial.
* Prior Therapy: Prior lines of anticancer therapy allowed as described in eligibility section above by disease status. Washout periods from prior therapy are as follows:

  * Myelosuppressive chemotherapy: Last dose given 14 days prior to enrollment.
  * Small molecule targeted therapies (anti-neoplastic agents including retinoids): Last dose given 7 days prior to enrollment.
  * Monoclonal antibodies: Last given at least 7 days or 3 half-lives, whichever is longer, prior to enrollment.
  * Radiation:

    * Craniospinal irradiation: Last fraction received minimum of six weeks prior to enrollment
    * All other radiation: Last fraction received minimum of 14 days prior to enrollment
  * Hematopoietic stem cell transplant: Date of autologous stem cell infusion following myeloablative chemotherapy must have been a minimum of 12 weeks prior to enrollment. Patients are not eligible post allogeneic stem cell transplant.
  * Cellular therapies (including CAR-T cells, NK cells, other related cellular therapies): 21 days from the last cellular therapy infusion prior to enrollment and recovery from all associated toxicities
  * 131I-MIBG therapy: Last therapy received a minimum of 6 weeks prior to enrollment.
* Age: Patients 1 - 30 years of age at the time of enrollment are eligible for this study.
* Performance level: Patients must demonstrate adequate performance level as measured by Karnofsky ≥ 70% for patients aged 16 years or older, OR Lansky ≥ 70% for patients younger than 16 years. Please see Appendix A for performance score measurement.
* Participants must meet the following organ and marrow function as defined below:
* Adequate bone marrow function as defined as BOTH of the following:

  * Peripheral absolute neutrophil count (ANC) ≥ 750/uL. Must be more than 14 days from last administration of long-acting myeloid stimulating factor (e.g. pegfilgrastim) or 7 days from last administration of short- acting myeloid stimulating factor (e.g. filgrastim or sargramostim)
  * Peripheral platelet count ≥ 75,000/uL. Must be without support, defined as at least 7 days from last platelet transfusion and/or platelet stimulating agent.
* Adequate renal function as defined as EITHER of the following:

  * Radioisotope GFR ≥ 70ml/min/1.73 m2
  * Serum creatinine based on age/sex as follows:
  * Age Maximum Serum Creatinine (mg/dL)

    * 1 to < 2 years Male 0.6 Female 0.6
    * 2 to < 6 years Male 0.8 Female 0.8
    * 6 to < 12 years Male 1.0 Female 1.0
    * 12 to < 13 years Male 1.2 Female 1.2
    * 13 to < 16 years Male 1.5 Female 1.4

      ---≥ 16 years Male 1.7 Female 1.4
    * The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR.
* Adequate liver function defined as ALL of the following:

  * Total bilirubin ≤ 1.5 x ULN for age*
  * ALT ≤ 3.0 x ULN for age (≤ 135 U/L). For the purpose of this study, the ULN for ALT is 45 U/L
  * Albumin > 3 g/dL --*If patient has known Gilbert syndrome, direct bilirubin should be used to measure liver function instead of total bilirubin. Direct bilirubin must be within normal limits for age for these patients.
* Adequate cardiac function measured by echocardiogram as defined as EITHER of the following:

  * Shortening fraction of ≥ 27%
  * Ejection fraction of ≥ 50%
* Adequate blood pressure as defined by BOTH of the following:

  * Patients must have < Grade 2 hypertension AND
  * Be on no more than one standing antihypertensive
* Adequate pulmonary function: Patients must have adequate pulmonary function, defined as:

  * No dyspnea at rest
  * No exercise intolerance
  * Room air O2 saturation >94%
  * Not on chronic oxygen therapy
* Adequate pancreatic function, defined as lipase < 1.5 x ULN
* Able to comply with protocol requirements
* Adequate contraception: The effects of naxitamab on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, participants with potential to become pregnant or to impregnate a partner must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a participant become pregnant or suspect they are pregnant while they or their partner is participating in this study, they should inform the treating physician immediately. Patients treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of protocol therapy.
* Ability to understand and/or the willingness of their parent or legally authorized representative to sign a written informed consent document.

Exclusion Criteria:

* Chronic (more than 2 weeks duration) diarrhea > grade 1
* Prior receipt of naxitamab
* Untreated central nervous system (CNS) metastatic disease
* Pregnant or currently breast feeding: Pregnant participants are excluded from this study because protocol therapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the parent with protocol therapy, participants planning to continue breastfeeding are excluded from the study.
* Clinically significant arrhythmias, i.e. those that cause clinical symptoms or require medications for control of symptoms
* Prior allergic reaction to irinotecan or temozolomide
* Discontinuation of prior irinotecan or temozolomide due to unacceptable toxicity
* Discontinuation of prior GD2 directed immunotherapy due to unacceptable toxicity other than allergic reaction
* Serious intercurrent illness
* Active uncontrolled infection
* Existing major organ dysfunction CTCAE >Grade 2, except for hearing loss and hematological status, kidney, and liver function as described in eligibility criteria
* Concomitant Medication Restrictions:

  * Patients may not be receiving immunosuppressive medications including pharmacologic doses of glucocorticoids or immunomodulatory agents due to concern for inhibition of antibody effect. Local and inhaled steroid agents are permitted.
  * Patients may not be receiving concurrent anti-cancer agents or radiotherapy.
  * Patients may not have received valproic acid within 14 days prior to enrollment.
  * Patients may not have received strong CYP3A4 inducers, strong CYP3A4 inhibitors, or strong UGT1A1 inhibitors within 14 days prior to enrollment.

    * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recommended duration of naxitamab infusion | Assessed at the end of the first cycle of treatment, where 1 cycle is 21 days
  The duration of naxitamab infusion that is safe and tolerable will be measured using the endpoint of an occurrence of any dose limiting toxicity. A modified 3+3 design will be used, where the 'modification' permits a single duration level de-escalation in addition to the typical duration group level escalation.

SECONDARY OUTCOMES:
Frequency of severe infusion related pain as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) | Assessed days 1 and 8 for Cycles 1 through 6, where 1 cycle is 21 days
  Frequency of CTCAE severe infusion related pain is defined as the count of all participants that experience a grade 3 or higher pain event as measured by CTCAE version 5.
Frequency of severe infusion related pain as measured by the Pediatric Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PEDS PRO-CTCAE) | Assessed days 1 and 8 for Cycles 1 through 6, where 1 cycle is 21 days
  Frequency of PEDS PRO-CTCAE severe infusion related pain is defined as the count of all participants that experience a score of 3 or greater on Question 1b of the PRO-CTCAE instrument.
Frequency of grade 3 or higher infusion related pain as measured by The Face, Legs, Activity, Cry, and Consolability (FLACC) Scale | Assessed on every naxitamab infusion day (days 1, 3, and 5) for both Cycle 1 and 2, where 1 cycle is 21 days
  Frequency of FLACC severe infusion related pain is defined as the count of all participants that experience a score of 7 or greater on the FLACC scale instrument.
Frequency of grade 3 or higher infusion related pain as measured by the Wong-Baker FACES scale | Assessed on every naxitamab infusion day (days 1, 3, and 5) for both Cycle 1 and 2, where 1 cycle is 21 days
  Frequency of FACES severe infusion related pain is defined as the count of all participants that experience a score of 4 or greater on the Wong-Baker FACES instrument.
Frequency of grade 3 or higher related pain as measured by the Numeric Rating Scale (NRS) | Assessed on every naxitamab infusion day (days 1, 3, and 5) for both Cycle 1 and 2, where 1 cycle is 21 days
  Frequency of NRS severe infusion related pain is defined as the count of all participants that experience a score of 7 or greater on the Numeric Rating Scale (NRS) instrument.
Frequency of additional infusion-related toxicity | Assessed at each clinic visit throughout the duration of treatment and for 35 days following the last dose of treatment, approximately 161 days
  Frequency of additional infusion-related toxicity will be defined as the count of toxicities which necessitate additional supportive care or interventions (i.e. an outpatient that requires hospital admission; an inpatient that requires ICU transfer).
Overall Best Response | Assessed at the end of 6 cycles of protocol chemoimmunotherapy, approximately 126 days
  Overall best response (as defined per International Neuroblastoma Response Committee criteria) at or before the end of 6 cycles of protocol chemoimmunotherapy.
Progression-Free Survival (PFS) | Assessed quarterly until withdrawal of consent or completion of the study (1 year follow-up after last treatment dose given to last enrolled patient).
  PFS time, defined as time from first response until first occurrence of relapse, progression, or death due to disease. Participants without an event will be censored at the time of last contact.
Overall Survival (OS) | Assessed quarterly until withdrawal of consent or completion of the study (1 year follow-up after last treatment dose given to last enrolled patient).
  OS time, defined as the time from first study treatment to death due to any cause, or censored at date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, MD, MS, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu